CLINICAL TRIAL: NCT02869022
Title: A Prospective, Randomized, Single Blind, Multicenter Phase III Study of Organ Perfusion With Custodiol-N Solution Compared With Custodiol Solution in Heart Transplantation
Brief Title: Study of Organ Perfusion With Custodiol-N Solution Compared With Custodiol Solution in Heart Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. F. Köhler Chemie GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL-N-HTX-CSM-III/04/12; 2012-001112-29 (EudraCT Number)
Record Dates: First submitted 2015-08-11; First posted 2016-08-16 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Custodiol-N solution; Heart Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Custodiol-N (Experimental): comparison of two perfusion solutions, Custodiol-N versus Custodiol, in heart transplantation
  Interventions: Drug: Custodiol-N; Procedure: organ perfusion for heart transplantation
- Custodiol (Active Comparator): comparison of two perfusion solutions, Custodiol-N versus Custodiol, in heart transplantation
  Interventions: Drug: Custodiol; Procedure: organ perfusion for heart transplantation

INTERVENTIONS:
Drug: Custodiol-N — comparison of two Solutions, Custodiol-N versus Custodiol, for organ Perfusion in heart transplantation
  Arms: Custodiol-N
Drug: Custodiol — comparison of two Solutions, Custodiol-N versus Custodiol, for organ Perfusion in heart transplantation
  Arms: Custodiol
Procedure: organ perfusion for heart transplantation

SUMMARY:
The objective of this investigation is to demonstrate non-inferiority in outcome of Custodiol-N against Custodiol in heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

Donor criteria:

* deceased donors should fulfil the criteria for organ donation (SCD) Patient criteria
* recipients awaiting their first transplant
* recipients ≥ 18 and >/= 65 years
* recipient's signed informed consent
* waiting list

Exclusion Criteria:

Donor criteria:

* not applicable

Patient criteria:

* recipients participating in another interventional study
* pregnant or lactating patients
* history/demonstration of HIV antibodies or AIDS
* multiorgan transplantation
* transMedics pump
* the explantation team is affiliated another clinic than transplantation team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Creatine kinase Myocard type "CK-MB" peak value | from 4 to 168 hours after release of the aortic cross clamp
  day 1: measurements 4, 8, 12, 16, 20, 24 hours ± 30 min; day 2-3: measurements 8, 16 and 24 hours ± 2 hours; day 4-7 one time/day

SECONDARY OUTCOMES:
Catecholamine requirement | from entry to the trial up to day 7
  defined as "yes" or "no"
Patient survival | at 7 days and 1, 3 and 12 months
Complications | from the time of the transplantation up to day 7
  occurrence, severity, type, and duration

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Szabo, Prof. Dr., Principal Investigator — Abt. Herzchirugie, Universitätsklinikum Heidelberg
Locations (9):
- Universitätsklinik für Chirurgie-Klin. Abteilung für Herzchirurgie, MUW-AKH Wien, Vienna, Austria
- Germany (8):
  - Klinik für Thorax- und Kardiovaskularchirurgie, Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Klinik für Herz-, Thorax- und Gefäßchirurgie, Deutsches Herzzentrum Berlin, Berlin
  - Klinik für Kardiovaskuläre Chirurgie, Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinik für Herz- und Gefäßchirurgie, Universitätszentrum Freiburg Bad Krotzingen, Freiburg im Breisgau
  - Klinik für Gefäßchirurgie, Universitäres Herzzentrum am UKE Hamburg, Hamburg
  - Abt. Herzchirugie, Universitätsklinikum Heidelberg, Heidelberg
  - Klinik für Herz- und Thoraxchirurgie, Universitätsklinikum Jena, Jena
  - Herz- Thorax- und herznahe Gefäßchirurgie, Klinikum der Universität Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: Undecided